CLINICAL TRIAL: NCT00595361
Title: The Effect of Beta-2 Adrenergic Polymorphisms on the Bronchoprotective Effects of Regular Salmeterol Treatment in Asthma
Brief Title: How Different Beta-2 Receptor Genotypes Affect an Asthmatic's Response to Regular Salmeterol Treatment
Acronym: SECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Director, Asthma Research Center, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-P-002199
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: asthma; exercise induced asthma; exercise induced bronchoconstriction; long acting beta agonist; salmeterol; exercise challenge; bronchoprotection; beta 2 adrenergic receptor polymorphisms; pharmacogenetics
MeSH Terms: conditions — Asthma; Asthma, Exercise-Induced | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arg/Arg (Active Comparator): Arg/Arg subjects on 2 week salmeterol treatment
  Interventions: Drug: salmeterol
- Gly/Gly (Active Comparator): Gly/Gly subjects on 2 week salmeterol treatment
  Interventions: Drug: salmeterol

INTERVENTIONS:
Drug: salmeterol — salmeterol 50 micrograms twice daily for 2 weeks

SUMMARY:
The purpose of the study is to find out how well a long-acting beta agonist like salmeterol works in people with different forms of the same gene. Our hypothesis is that asthmatics with the Arg/Arg genotype will have loss of bronchoprotection against exercise-induced asthma with regular salmeterol treatment, as compared to asthmatics with the Gly/Gly genotype.

DETAILED DESCRIPTION:
In many patients with asthma, exercise-induced bronchoconstriction is a common and oftentimes limiting characteristic. Inhaled β2-adrenoreceptor agonists like albuterol are the most effective treatments available for the relief of acute asthma symptoms. However, there is evidence that regular use may lead to adverse effects in some patients. Previous studies have shown that polymorphisms of the β2-adrenergic receptor can influence airway responses to regular inhaled beta-agonist treatment.

Pharmacogenetics is the study of how genetic differences influence the variability in patients' responses to therapy, both therapeutic and adverse. Genetic susceptibility and environmental factors both play major roles in the etiology of asthma. The strong familial clustering of asthma has lead to a surge of research into the genetic predisposition of asthma. The aim of the present study is to utilize a double-blinded prospective cohort study to investigate whether genotype-specific effects occur when assessing the duration of protection conferred against exercise-induced bronchoconstriction by regular salmeterol treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* 18 to 50 years of age
* Resting FEV1 ≥ 65% of predicted normal
* Exercise-induced bronchoconstriction defined as a decrease in FEV1 of ≥ 20% following a standardized exercise challenge when compared to pre-exercise baseline FEV1 value measured 5 minutes before exercise
* Must be Arg/Arg or Gly/Gly genotype

Exclusion Criteria:

* Long-acting beta agonist use within 12 weeks of the first exercise challenge
* Smoking within past 12 months
* Greater than 10-pack years smoking history
* Unresolved signs and/or symptoms of an upper respiratory tract infection within 4 weeks of first exercise challenge
* Asthma exacerbation within 4 weeks of first exercise challenge requiring change in type, dose or frequency of medications and/or an unscheduled visit to an health care provider, including emergency room or hospital
* Subject has exercised or performed strenuous activity within 72 hours of the first exercise challenge
* Subject has been exposed to cold air sufficient to provoke symptoms of bronchospasm within 2 hours of exercise challenge
* In addition to asthma, the subject has an active, acute or chronic pulmonary disorder documented by history, physical examination, or chest x-ray
* Subject has evidence of ischemic, valvular, hypertrophic, familial or other forms of heart disease that would put the subject at risk during exercise testing or that would interfere with the ability to achieve protocol-specified heart rates during exercise testing
* Subject has used systemic corticosteroids within 1 month of first exercise challenge

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, M.D., Principal Investigator — Asthma Research Center, Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Israel E, Drazen JM, Liggett SB, Boushey HA, Cherniack RM, Chinchilli VM, Cooper DM, Fahy JV, Fish JE, Ford JG, Kraft M, Kunselman S, Lazarus SC, Lemanske RF, Martin RJ, McLean DE, Peters SP, Silverman EK, Sorkness CA, Szefler SJ, Weiss ST, Yandava CN. The effect of polymorphisms of the beta(2)-adrenergic receptor on the response to regular use of albuterol in asthma. Am J Respir Crit Care Med. 2000 Jul;162(1):75-80. doi: 10.1164/ajrccm.162.1.9907092. PMID 10903223
- [Result] Israel E, Chinchilli VM, Ford JG, Boushey HA, Cherniack R, Craig TJ, Deykin A, Fagan JK, Fahy JV, Fish J, Kraft M, Kunselman SJ, Lazarus SC, Lemanske RF Jr, Liggett SB, Martin RJ, Mitra N, Peters SP, Silverman E, Sorkness CA, Szefler SJ, Wechsler ME, Weiss ST, Drazen JM; National Heart, Lung, and Blood Institute's Asthma Clinical Research Network. Use of regularly scheduled albuterol treatment in asthma: genotype-stratified, randomised, placebo-controlled cross-over trial. Lancet. 2004 Oct 23-29;364(9444):1505-12. doi: 10.1016/S0140-6736(04)17273-5. PMID 15500895
- [Result] Wechsler ME, Lehman E, Lazarus SC, Lemanske RF Jr, Boushey HA, Deykin A, Fahy JV, Sorkness CA, Chinchilli VM, Craig TJ, DiMango E, Kraft M, Leone F, Martin RJ, Peters SP, Szefler SJ, Liu W, Israel E; National Heart, Lung, and Blood Institute's Asthma Clinical Research Network. beta-Adrenergic receptor polymorphisms and response to salmeterol. Am J Respir Crit Care Med. 2006 Mar 1;173(5):519-26. doi: 10.1164/rccm.200509-1519OC. Epub 2005 Dec 1. PMID 16322642
- [Result] Ramage L, Lipworth BJ, Ingram CG, Cree IA, Dhillon DP. Reduced protection against exercise induced bronchoconstriction after chronic dosing with salmeterol. Respir Med. 1994 May;88(5):363-8. doi: 10.1016/0954-6111(94)90042-6. PMID 7913549
- [Result] Yates DH, Worsdell M, Barnes PJ. Effect of regular salmeterol treatment on albuterol-induced bronchoprotection in mild asthma. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):988-91. doi: 10.1164/ajrccm.156.3.9610051. PMID 9310023
- [Result] Nelson JA, Strauss L, Skowronski M, Ciufo R, Novak R, McFadden ER Jr. Effect of long-term salmeterol treatment on exercise-induced asthma. N Engl J Med. 1998 Jul 16;339(3):141-6. doi: 10.1056/NEJM199807163390301. PMID 9664089
- [Result] Palmer CN, Lipworth BJ, Lee S, Ismail T, Macgregor DF, Mukhopadhyay S. Arginine-16 beta2 adrenoceptor genotype predisposes to exacerbations in young asthmatics taking regular salmeterol. Thorax. 2006 Nov;61(11):940-4. doi: 10.1136/thx.2006.059386. Epub 2006 Jun 13. PMID 16772309
- [Result] Israel E. Genetics and the variability of treatment response in asthma. J Allergy Clin Immunol. 2005 Apr;115(4 Suppl):S532-8. doi: 10.1016/j.jaci.2005.01.029. PMID 15806036
- [Derived] Bonini M, Permaul P, Kulkarni T, Kazani S, Segal A, Sorkness CA, Wechsler ME, Israel E. Loss of salmeterol bronchoprotection against exercise in relation to ADRB2 Arg16Gly polymorphism and exhaled nitric oxide. Am J Respir Crit Care Med. 2013 Dec 15;188(12):1407-12. doi: 10.1164/rccm.201307-1323OC. PMID 24228710

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arg/Arg | Gly/Gly
Started | 12 | 18
Completed | 12 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arg/Arg | Gly/Gly | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (2.4) | 27.2 (1.4) | 26.6 (1.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Maximum Percent Fall in FEV1 After Exercise Challenge at the End of the 2-week Treatment Period Between Arg/Arg and Gly/Gly Patients
Time Frame: 2 weeks after exercise challenge
Measure: Mean (Standard Deviation); unit: % fall FEV1
Arm/Group | Arg/Arg | Gly/Gly
Number analyzed (Participants) | 12 | 14
% fall FEV1 | 12.6 (4.5) | 16.5 (2.9)

2. Secondary Outcome: Comparison of the Maximum Percent Fall in FEV1 From Pre-salmeterol Baseline to the End of the 2-week Treatment Period Between Arg/Arg and Gly/Gly Patients
Time Frame: 2 weeks from pre-salmeterol baseline
Measure: Mean (Standard Deviation); unit: % fall FEV1
Arm/Group | Arg/Arg | Gly/Gly
Number analyzed (Participants) | 12 | 14
% fall FEV1 | 5.9 (19.9) | 4.3 (10.6)

3. Secondary Outcome: Comparison of the Maximum Percent Fall in FEV1 After 1st Dose of Salmeterol to the End of the 2-week Treatment Period Between Arg/Arg and Gly/Gly Subjects
Time Frame: 2 weeks after 1st dose of Salmeterol
Measure: Mean (Standard Deviation); unit: % fall FEV1
Arm/Group | Arg/Arg | Gly/Gly
Number analyzed (Participants) | 12 | 14
% fall FEV1 | -12.6 (17.1) | -16.5 (10.9)

ADVERSE EVENTS:
Arm/Group | Arg/Arg | Gly/Gly
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No